CLINICAL TRIAL: NCT05324865
Title: The Effect of Progressive Muscle Relaxation on Psychological Symptoms and Mental Well-Being in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Omer Tanriverdi, Nursing, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hasan kalyoncu University Omer
Record Dates: First submitted 2022-01-10; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenic Psychoses
Keywords: Schizophrenic; relaxation exercise; nursing; psychological symptoms
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Information about the experimental group was given. Progressive muscle relaxation (PMR) for 6 weeks to patients with schizophrenia will be heard. At the end of 6 weeks, psychiatric evaluation and mental well-being scale will be used.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Control Group (No Intervention): Patient identification form, psychological evaluation form and mental health form were filled in for the control group. At the end of 6 weeks, the psychological evaluation form and the mental well-being form were filled again without any intervention.

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation PMR is a technique that provides relaxation in the whole body by voluntary and regular relaxation of large muscle groups in the human body, which is included in mind-body applications.
  Arms: Experimental Group

SUMMARY:
Schizophrenia is a mental illness that progresses with delusions or hallucinations, causes changes in interpersonal communication, thoughts and behaviors, continues with recovery and repetitions, and in which the interpretation of reality is impaired. Drug treatment alone is not sufficient in schizophrenia, and it is known that negative symptoms continue even in patients with a good response to drug treatment. For this reason, complementary therapies, psychosocial approaches and rehabilitation in addition to drug therapy increase the effectiveness of the treatment.

DETAILED DESCRIPTION:
Schizophrenia is a mental illness that progresses with delusions or hallucinations, causes changes in interpersonal communication, thoughts and behaviors, continues with recovery and repetitions, and in which the interpretation of reality is impaired. Drug treatment alone is not sufficient in schizophrenia, and it is known that negative symptoms continue even in patients with a good response to drug treatment. For this reason, complementary therapies, psychosocial approaches and rehabilitation in addition to drug therapy increase the effectiveness of the treatment.It is seen that the tension, the effects of stress, the state of anxiety, blood pressure, heart rate, lactic acid production, sensitivity to pain are reduced by performing relaxation exercises in a suitable environment, regularly and in accordance with the technique. Helps you think positively Studies involving patients with schizophrenia have also proven the beneficial effect of progressive relaxation, with positive changes observed through relieving anxiety, reducing psychological stress, and increasing psychological well-being.

ELIGIBILITY:
Inclusion Criteria:• Being 18 years or older,

* Having a confirmed diagnosis of schizophrenia for at least 6 months
* Having the ability to communicate and read,
* Volunteering to participate in the research.

Exclusion Criteria:• Being closed to communication,

* Not complying with the principle of voluntarism
* Patients in acute exacerbation period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 10 minute
  Patients' personal information (age, gender, marital status, educational status, income status, employment status) and disease information (year of disease onset, is the drug treatment sufficient, does the drug take the drug regularly, is there a regular check-up, is there any substance addiction) (cigarette, alcohol), are there any non-drug treatment methods in the fight against the disease) constitute questions.
Warwick-Edinburgh Mental Well-Being Scale | 15 minute
  The scale consists of 14 positive items and has a 5-point Likert-type answer key. High scores from the scale indicate high mental well-being.
Psychiatric Rating Scale(PRS) | 15 minute
  This form consists of 18 items. The items of the scale are scored between 0-6. It shows that the severity of the disease increases as the scoring increases.